CLINICAL TRIAL: NCT02332863
Title: Comparison of Traditional Back-loaded Fiducial Needles With Preloaded Fiducial Needles in EUS-guided Fiducial Marker Placement for Image-guided Radiation Therapy in Patients With Pancreatic Cancer: A Multicenter Randomized Controlled Trial.
Brief Title: Comparison of Back-loaded vs Preloaded Fiducial Needles in EUS-guided Fiducial Marker Placement in Pancreatic Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-1711.cc
Record Dates: First submitted 2014-09-22; First posted 2015-01-07 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Image guided radiation therapy; Fiducial marker placement; Endoscopic ultrasound
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Back-loaded needle (Active Comparator): The patients will undergo Linear EUS and have fiducial marker placement via a traditional 22G back-loaded needle. CRFs will be used to record data for primary and secondary endpoints.
  Interventions: Device: Back-loaded Needle (Device)
- Preloaded Needle (Experimental): The patients will undergo Linear EUS and have fiducial marker placement via a traditional 22G preloaded needle. CRFs will be used to record data for primary and secondary endpoints.
  Interventions: Device: Preloaded Needle (Device)

INTERVENTIONS:
Device: Back-loaded Needle (Device) — Fiducial marker placement via a traditional 22G back-loaded needle will be performed with multiple endpoints recorded:
  * total length of procedure
  * how many markers are successfully deployed
  * technical success
  Fiducial marker location will be confirmed via fluoroscopy at time of placement and on 4D treatment planning CT ordered by the radiation oncologist for simulation.
  Arms: Back-loaded needle
Device: Preloaded Needle (Device) — Fiducial marker placement via a novel 22G preloaded needle will be performed with multiple endpoints recorded:
  * total length of procedure
  * how many markers are successfully deployed
  * technical success
  Fiducial marker location will be confirmed via fluoroscopy at time of placement and on 4D treatment planning CT ordered by the radiation oncologist for simulation.
  Arms: Preloaded Needle

SUMMARY:
Endoscopic ultrasound (EUS) has been pivotal in accomplishing image guided radiation therapy (IGRT) in patients with pancreatic cancer by allowing precise contouring and identification of target lesions in the pancreas via placement of fiducials using fine needle aspiration (FNA) needles. Currently, back-loading the fiducials is the only option for preparing delivery of fiducials via the EUS approach. A prototype 22-Gauge EUS needle preloaded with four fiducials has recently been developed, and used in a porcine models with successful results. There are no randomized controlled trials comparing total duration of time needed for placement of fiducials using technical success of the traditional back- loading technique of fiducial markers to the new preloaded needles in regards to EUS based fiducial marker placement for IGRT in pancreatic cancer.

Hypotheses

Use of a 22 G preloaded needle for EUS guided fiducial marker placement in patients with pancreatic cancer will:

1. Be delivered in at least require 60% less of the procedure time that it takes for traditional back-loaded 22G needles
2. Improve overall procedure efficiency
3. Maintain comparable technical success and adverse event rates.

Primary Aims

1) To compare the procedure time of 22G needle placement of three Visicoil (brand of flexible linear back-loaded fiducial markers) fiducial markers and 22G needle preloaded fiducial markers.

Secondary Aims

1. To compare adverse event rates in 22G needle placement of Visicoil fiducial markers and 22G needle preloaded fiducial markers
2. To compare endpoints of technical success defined as proper placement of two to three fiducial markers in a pancreatic neoplasm in 22G needle placement of Visicoil fiducial markers and 22G needle preloaded fiducial markers.

DETAILED DESCRIPTION:
Pancreatic cancer is the twelfth most common cancer worldwide. Neoadjuvant chemoradiation therapy in patients with borderline resectable pancreatic adenocarcinoma has become standard of care and is associated with higher rates of complete resection ultimately with improvement of overall survival in this patient population. Radiation therapy to a soft tissue organ such as the pancreas can be difficult, as it is not readily visualized radiographically. Image guided radiation therapy (IGRT) is a commonly implemented modality for delivering high doses of radiation directed at cancer tissue, while reducing collateral damage to adjacent healthy tissue. Fiducials, which are inert radiographic markers typically made from gold or carbon, can be placed in and around the tumor to delineate tumor margins to allow for IGRT Endoscopic ultrasound (EUS) has been pivotal in accomplishing IGRT by allowing precise contouring and identification of target lesions in the pancreas via placement of fiducials. This has traditionally been accomplished with the use of 19-gauge or 22-gauge fine needle aspiration (FNA) needles. To prepare the needle for fiducial placement, one to two fiducials are manually back-loaded into the tip of the needle after the stylet has been removed. In order to hold the fiducials within the needle, sterile lubrication or bone wax can be applied. Once the pancreatic mass has been targeted, fiducial injection can be accomplished via stylet reinsertion or sterile water injection. Currently, back-loading the fiducials is the only option for preparing delivery of fiducials via the EUS approach. Difficulties associated with fiducial loading and deployment can increase procedure duration due to cumbersome fiducial back-loading, fiducial misplacement & migration, as well as inability to pass the fiducial marker through the needle due to endoscope angulation. Observational studies have sited a technical success rate of 86-100% using 19 and/or 22 gauge needles with average procedure time between 7-12 minutes using the fiducial back-loading technique.

A new mode of fiducial delivery has recently been developed that hopes to circumvent some of the technical issues inherent to traditional fiducial marker loading and deployment. A prototype 22-Gauge EUS needle preloaded with four fiducials has been used in a porcine models with successful deployment 95.6% of the time all accurate on predetermined targets. They were deemed easy to pass, relatively easy to deploy, and easily visualized on EUS, with excellent fluoroscopic and CT visualization. In addition, time for deployment was on average less than 60 seconds.

To date, there is no randomized controlled trials comparing total duration of time needed for placement of fiducials using technical success of the traditional back- loading technique of fiducial markers to the new preloaded needles in regards to EUS based fiducial marker placement for IGRT in pancreatic cancer.

This will be a multicenter randomized controlled trial. Randomization be performed and patients will undergo Linear EUS and have fiducial marker placement via a traditional 22G back-loaded needle (Visicoil) or the new 22G preloaded needle (PreLoad4). Multiple endpoints will be recorded, including total length of procedure, how many markers are successfully deployed, and technical success (Ease of passage of delivery system, ease of deployment of fiducials, EUS visualization of delivery system needle, EUS visual appearance of fiducials, and time for fiducial placement defined as starting at time of removing the needle from its packaging and ending time as removal of needle after final marker deployment). Fiducial marker location will be confirmed via fluoroscopy at time of placement and on 4D treatment planning CT ordered by the radiation oncologist for simulation. Patients will be discharged home after post procedure recovery. Patients will be contacted at home by a research coordinator or endoscopy staff 24-48 hours and 7-10 days after the procedure to document any immediate and delayed complications. Patients will return for their IGRT visit, and any evidence of fiducial marker migration will be recorded by the radiation oncologist.

Hypotheses

Use of a 22 G preloaded needle for EUS guided fiducial marker placement in patients with pancreatic cancer will:

1. Be delivered in at least require 60% less of the procedure time that it takes for traditional back-loaded 22G needles
2. Improve overall procedure efficiency
3. Maintain comparable technical success and adverse event rates.

Primary Aims

1) To compare the procedure time of 22G needle placement of three Visicoil fiducial markers and 22G needle preloaded fiducial markers.

Secondary Aims

1. To compare adverse event rates in 22G needle placement of Visicoil fiducial markers and 22G needle preloaded fiducial markers
2. To compare endpoints of technical success defined as proper placement of two to three fiducial markers in a pancreatic neoplasm in 22G needle placement of Visicoil fiducial markers and 22G needle preloaded fiducial markers.

ELIGIBILITY:
Inclusion Criteria:

• Patients with pathologically confirmed pancreatic cancer referred for image guided radiation therapy (IGRT)

Exclusion Criteria:

* Age <18
* Inability to consent
* Known coagulopathy/thrombocytopenia (INR >1.5, platelets <75)
* Patients on antiplatelet/anticoagulant medication that cannot safely be discontinued 5-7 days prior to the procedure
* Gold allergy
* Current infection
* EUS evidence of vessel interfering with path of fiducial marker
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Wani, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida

REFERENCES:
- [Background] Colbert LE, Hall WA, Nickleach D, Switchenko J, Kooby DA, Liu Y, Gillespie T, Lipscomb J, Kauh J, Landry JC. Chemoradiation therapy sequencing for resected pancreatic adenocarcinoma in the National Cancer Data Base. Cancer. 2014 Feb 15;120(4):499-506. doi: 10.1002/cncr.28530. Epub 2014 Jan 3. PMID 24390739
- [Background] Fuss M, Wong A, Fuller CD, Salter BJ, Fuss C, Thomas CR. Image-guided intensity-modulated radiotherapy for pancreatic carcinoma. Gastrointest Cancer Res. 2007 Jan;1(1):2-11. PMID 19262697
- [Background] Reese AS, Lu W, Regine WF. Utilization of intensity-modulated radiation therapy and image-guided radiation therapy in pancreatic cancer: is it beneficial? Semin Radiat Oncol. 2014 Apr;24(2):132-9. doi: 10.1016/j.semradonc.2013.11.003. PMID 24635870
- [Background] Javed S, Bhutani MS. Endoscopic ultrasound-guided radiation therapy in pancreatic cancer. Minerva Gastroenterol Dietol. 2013 Dec;59(4):377-86. PMID 24212355
- [Background] Kooby DA, Gillespie TW, Liu Y, Byrd-Sellers J, Landry J, Bian J, Lipscomb J. Impact of adjuvant radiotherapy on survival after pancreatic cancer resection: an appraisal of data from the national cancer data base. Ann Surg Oncol. 2013 Oct;20(11):3634-42. doi: 10.1245/s10434-013-3047-x. Epub 2013 Jun 15. PMID 23771249
- [Background] Suzuki R, Irisawa A, Bhutani MS. Endoscopic ultrasound-guided oncologic therapy for pancreatic cancer. Diagn Ther Endosc. 2013;2013:157581. doi: 10.1155/2013/157581. Epub 2013 Feb 24. PMID 23533319
- [Background] Khashab MA, Kim KJ, Tryggestad EJ, Wild AT, Roland T, Singh VK, Lennon AM, Shin EJ, Ziegler MA, Sharaiha RZ, Canto MI, Herman JM. Comparative analysis of traditional and coiled fiducials implanted during EUS for pancreatic cancer patients receiving stereotactic body radiation therapy. Gastrointest Endosc. 2012 Nov;76(5):962-71. doi: 10.1016/j.gie.2012.07.006. PMID 23078921
- [Background] Ammar T, Cote GA, Creach KM, Kohlmeier C, Parikh PJ, Azar RR. Fiducial placement for stereotactic radiation by using EUS: feasibility when using a marker compatible with a standard 22-gauge needle. Gastrointest Endosc. 2010 Mar;71(3):630-3. doi: 10.1016/j.gie.2009.11.023. PMID 20189527
- [Background] Park WG, Yan BM, Schellenberg D, Kim J, Chang DT, Koong A, Patalano C, Van Dam J. EUS-guided gold fiducial insertion for image-guided radiation therapy of pancreatic cancer: 50 successful cases without fluoroscopy. Gastrointest Endosc. 2010 Mar;71(3):513-8. doi: 10.1016/j.gie.2009.10.030. PMID 20189509
- [Background] Davila Fajardo R, Lekkerkerker SJ, van der Horst A, Lens E, Bergman JJ, Fockens P, Bel A, van Hooft JE. EUS-guided fiducial markers placement with a 22-gauge needle for image-guided radiation therapy in pancreatic cancer. Gastrointest Endosc. 2014 May;79(5):851-5. doi: 10.1016/j.gie.2013.12.027. Epub 2014 Feb 8. No abstract available. PMID 24518121
- [Background] DiMaio CJ, Nagula S, Goodman KA, Ho AY, Markowitz AJ, Schattner MA, Gerdes H. EUS-guided fiducial placement for image-guided radiation therapy in GI malignancies by using a 22-gauge needle (with videos). Gastrointest Endosc. 2010 Jun;71(7):1204-10. doi: 10.1016/j.gie.2010.01.003. PMID 20598247
- [Background] Owens DJ, Savides TJ. EUS placement of metal fiducials by using a backloaded technique with bone wax seal. Gastrointest Endosc. 2009 Apr;69(4):972-3. doi: 10.1016/j.gie.2008.05.052. Epub 2009 Jan 18. No abstract available. PMID 19152903
- [Background] Khara HS, Pineda-Bonilla JJ, Chaput KJ, Johal AS. Endoscopic ultrasound-guided placement of fiducial markers using a novel "wet-fill technique" without a bone wax seal. Endoscopy. 2013;45 Suppl 2 UCTN:E426-7. doi: 10.1055/s-0033-1358809. Epub 2013 Dec 13. No abstract available. PMID 24338173
- [Background] Pishvaian AC, Collins B, Gagnon G, Ahlawat S, Haddad NG. EUS-guided fiducial placement for CyberKnife radiotherapy of mediastinal and abdominal malignancies. Gastrointest Endosc. 2006 Sep;64(3):412-7. doi: 10.1016/j.gie.2006.01.048. PMID 16923491
- [Background] Varadarajulu S, Trevino JM, Shen S, Jacob R. The use of endoscopic ultrasound-guided gold markers in image-guided radiation therapy of pancreatic cancers: a case series. Endoscopy. 2010 May;42(5):423-5. doi: 10.1055/s-0029-1243989. Epub 2010 Mar 15. PMID 20232282
- [Background] Sanders MK, Moser AJ, Khalid A, Fasanella KE, Zeh HJ, Burton S, McGrath K. EUS-guided fiducial placement for stereotactic body radiotherapy in locally advanced and recurrent pancreatic cancer. Gastrointest Endosc. 2010 Jun;71(7):1178-84. doi: 10.1016/j.gie.2009.12.020. Epub 2010 Apr 1. PMID 20362284
- [Background] Draganov PV, Chavalitdhamrong D, Wagh MS. Evaluation of a new endoscopic ultrasound-guided multi-fiducial delivery system: a prospective non-survival study in a live porcine model. Dig Endosc. 2013 Nov;25(6):615-21. doi: 10.1111/den.12046. Epub 2013 Mar 12. PMID 23489989
- [Background] Fuccio L, Guido A, Larghi A, Antonini F, Lami G, Fabbri C. The role of endoscopic ultrasound in the radiation treatment of pancreatic tumor. Expert Rev Gastroenterol Hepatol. 2014 Sep;8(7):793-802. doi: 10.1586/17474124.2014.913479. Epub 2014 Apr 28. PMID 24766230
- [Derived] Machicado JD, Obuch JC, Goodman KA, Schefter TE, Frakes J, Hoffe S, Latifi K, Simon VC, Santangelo T, Ezekwe E, Edmundowicz SA, Brauer BC, Shah RJ, Hammad HT, Wagh MS, Attwell A, Han S, Klapman J, Wani S. Endoscopic Ultrasound Placement of Preloaded Fiducial Markers Shortens Procedure Time Compared to Back-Loaded Markers. Clin Gastroenterol Hepatol. 2019 Dec;17(13):2749-2758.e2. doi: 10.1016/j.cgh.2019.04.046. Epub 2019 Apr 28. PMID 31042578

RESULTS

PARTICIPANT FLOW:
Groups:
- Back-loaded Needle: The patients will undergo Linear EUS and have fiducial marker placement via a traditional 22G back-loaded needle. CRFs will be used to record data for primary and secondary endpoints.
  Back-loaded Needle (Device): Fiducial marker placement via a traditional 22G back-loaded needle will be performed with multiple endpoints recorded:
  * total length of procedure
  * how many markers are successfully deployed
  * technical success
  Fiducial marker location will be confirmed via fluoroscopy at time of placement and on 4D treatment planning CT ordered by the radiation oncologist for simulation.
- Preloaded Needle: The patients will undergo Linear EUS and have fiducial marker placement via a traditional 22G preloaded needle. CRFs will be used to record data for primary and secondary endpoints.
  Preloaded Needle (Device): Fiducial marker placement via a novel 22G preloaded needle will be performed with multiple endpoints recorded:
  * total length of procedure
  * how many markers are successfully deployed
  * technical success
  Fiducial marker location will be confirmed via fluoroscopy at time of placement and on 4D treatment planning CT ordered by the radiation oncologist for simulation.
Period: Overall Study
Arm/Group | Back-loaded Needle | Preloaded Needle
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Back-loaded Needle | Preloaded Needle | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 12 | 14 | 26
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [59 to 74] | 67 [59 to 75] | 66 [59 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 21 | 39
  Black | 2 | 0 | 2
  Hispanic | 2 | 0 | 2
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.8 (6.3) | 23.6 (4.2) | 24.7 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Procedure Duration Required for Placing the Fiducial Markers
Description: Duration of procedure for placing fiducial markers including: Fiducial package was opened start time (start stop watch) + Fiducial placement end time (end stop watch) = Placing Fiducial Markers Time
Time Frame: During scheduled procedure (approximately 1 hour)
Measure: Median (Inter-Quartile Range); unit: mintues
Arm/Group | Back-loaded Needle | Preloaded Needle
Number analyzed (Participants) | 22 | 22
mintues | 16 [12 to 24] | 9 [6 to 12]

2. Secondary Outcome: Total Procedure Time
Description: Total procedure time will be recorded during the procedure using a case report form (CRF) for Procedure Time
Time Frame: During scheduled procedure (approximately 1 hour)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Back-loaded Needle | Preloaded Needle
Number analyzed (Participants) | 22 | 22
minutes | 27 [23 to 28] | 25 [18 to 36]

3. Secondary Outcome: Number of Participants With Technical Success EUS Needle Visualization
Description: EUS needle visualization during the procedure will be recorded on a CRF for Scale of Technical Success.
Time Frame: During scheduled procedure (approximately 1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | Back-loaded Needle | Preloaded Needle
Number analyzed (Participants) | 22 | 22
Participants | 16 | 14

4. Secondary Outcome: Technical Success
Description: Defined as the proper placement of 3 fiducial markers in a pancreatic neoplasm in 2 different planes
Time Frame: During scheduled procedure (approximately 1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | Back-loaded Needle | Preloaded Needle
Number analyzed (Participants) | 22 | 22
Participants | 22 | 20

5. Secondary Outcome: Number of Participants With Visualization of Fiducials as Assessed by Radiation Oncology
Description: Fiducial location on CT scan will be assessed at patient's radiation oncology appointments for IGRT.
Time Frame: Several hours to 7 days after fiducial marker deployment
Measure: Count of Participants; unit: Participants
Arm/Group | Back-loaded Needle | Preloaded Needle
Number analyzed (Participants) | 22 | 22
Participants | 20 | 19

6. Secondary Outcome: Number of Participants With Inadvertent Deployment of Fiducials
Description: Whether inadvertent deployment of fiducials occurs will be recorded on a CRF for Data Acquisition
Time Frame: During scheduled procedure (approximately 1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | Back-loaded Needle | Preloaded Needle
Number analyzed (Participants) | 22 | 22
Participants | 1 | 1

7. Secondary Outcome: Number of Participants With Ease of Passage of Delivery System
Description: Ease of needle device passage through EUS will be recorded on a CRF form for technical success.
Time Frame: During scheduled procedure (approximately 1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | Back-loaded Needle | Preloaded Needle
Number analyzed (Participants) | 22 | 22
Participants
  Easy/minimal difficulty | 21 | 15
  Moderate/significant difficulty | 1 | 6
  Unable to pass needle | 0 | 1

8. Secondary Outcome: Number of Fiducials Placed
Description: Number of fiducials placed will be recorded during the procedure using a case report form (CRF) for Fiducial Placement Data
Time Frame: During scheduled procedure (about 90 minutes)
Measure: Median (Inter-Quartile Range); unit: fiducials
Arm/Group | Back-loaded Needle | Preloaded Needle
Number analyzed (Participants) | 22 | 22
fiducials | 3 [3 to 4] | 3 [3 to 4]

ADVERSE EVENTS:
Time Frame: Immediately after the procedure 24-48 hours after the procedure 7-10 days after the procedure
Description: Study coordinators assessed for procedure-related AEs immediately after, 24-48 hours, and at 5-7 days, with a structured questionnaire. AEs at 24-48 hours and at 5-7 days were assessed through a telephone call.
Arm/Group | Back-loaded Needle | Preloaded Needle
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 19/22 | 16/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Back-loaded Needle (N=22) | Preloaded Needle (N=22)
Abdominal Pain (Gastrointestinal disorders) | 11 | 8
Nausea and/or vomiting (Gastrointestinal disorders) | 6 | 3
Other (Gastrointestinal disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT02332863/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT02332863/SAP_001.pdf
  • Informed Consent Form (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT02332863/ICF_002.pdf